CLINICAL TRIAL: NCT00319735
Title: A Pilot Study With Cetuximab and Radiation Therapy for Patients With Surgically Resectable Esophageal and GE Junction Carcinomas: Hoosier Oncology Group Study (GI05-92)
Brief Title: Cetuximab and Radiation Therapy for Surgically Resectable Esophageal and Gastroesophageal (GE) Junction Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nasser Hanna, M.D. (Other)
Collaborators: Bristol-Myers Squibb (Industry); Walther Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Nasser Hanna, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG GI05-92
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy; Surgical Procedures, Operative; Histocompatibility Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational Treatment (Experimental): * Cetuximab 400 mg/m2 IV over 120 minutes Day -14 (Loading Dose)
  * Cetuximab 250 mg/m2 IV over 60 minutes Day -7
  * Cetuximab 250 mg/m2 IV over 60 minutes Days 1, 8, 15, 22, 29 and 36
  * Combined with radiation therapy for six weeks.
  * Surgery for esophageal resection after 6 to 8 week rest period.
  Subjects who consent will provide tissue samples.
  Interventions: Procedure: Radiation Therapy; Procedure: Surgery; Procedure: Tissue Sample

INTERVENTIONS:
Procedure: Radiation Therapy — External beam radiation therapy, beginning on day 1, 4500 cGy to esophagus with boost of 540 cGy at 180 cGy per fraction for 6 weeks
Procedure: Surgery — Surgical resection of primary tumor and adjacent mediastinal and/or celiac lymph nodes by a transthoracic approach after satisfactory hematologic and functional recovery within 8 weeks of completion of radiation therapy
Procedure: Tissue Sample — For patients who give their consent, fresh frozen tissue will be obtained per EUS at baseline, per EUS 2 weeks after the initiation of chemotherapy, and at the time of surgery for pathology submission

SUMMARY:
The interaction of epidermal growth factor receptor (EGFR) inhibitory agents such as cetuximab combined with radiation shows promising results. EGFR inhibitory agents also enhance radiation-induced apoptosis and inhibit radiation induced damage repair. These interactions may represent the principle effects that contribute to the synergy between EGFR and radiation.

This trial will investigate the feasibility and activity of this combination in patients with surgically resectable disease.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Cetuximab 400 mg/m2 IV over 120 minutes Day -14 (Loading Dose)
* Cetuximab 250 mg/m2 IV over 60 minutes, day -7.
* Cetuximab 250 mg/m2 IV over 60 minutes, days 1, 8, 15, 22, 29 and 36.
* External beam radiation therapy, beginning on day 1, 4500 cGy to esophagus with boost of 540 cGy at 180 cGy per fraction for 6 weeks.
* Surgical resection of primary tumor and adjacent mediastinal and/or celiac lymph nodes by a transthoracic approach after satisfactory hematologic and functional recovery within 8 weeks of completion of radiation therapy.
* For patients who give their consent, fresh frozen tissue will be obtained per EUS at baseline, per EUS 2 weeks after the initiation of cetuximab, and at the time of surgery for pathology submission.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of either squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction.
* Clinical stage IIA, IIB or III without metastatic disease
* Patients must have documented EGFR status or have tumor tissue available for assessment of EGFR status by IHC
* Patients must be surgical candidates as determined by surgical consult.
* Patients must agree to surgery.
* ECOG performance status 0 or 2
* Absolute neutrophil count (ANC) > 1,000 mm3
* Platelet count > 75,000 mm3· Hemoglobin > 10g/dL
* Bilirubin < 2.5 X upper limit of normal
* AST (SGOT) or ALT (SGPT) < 5.0 ´ upper limit of normal
* Creatinine < 2.0 X upper limit of normal

Exclusion Criteria:

* No history of or current brain metastasis.
* No significant history of uncontrolled cardiac disease; i.e. uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* No history of interstitial pneumonitis or pulmonary fibrosis, or suspicion of interstitial pneumonitis or pulmonary fibrosis on imaging.
* No concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).
* No prior use of radiation or chemotherapy for cancer of the esophagus or GE junction
* No prior therapy that specifically and directly targets the EGFR pathway (such as kinase inhibitors and antibodies directed against the HER family receptors).
* No prior severe infusion reaction to a monoclonal antibody.
* No major surgery within 28 days prior to being registered for protocol therapy.
* No clinically significant infections as judged by the treating investigator.
* No acute hepatitis or known HIV.
* No other active malignancies.
* Negative pregnancy test.
* No female patients currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Becerra, M.D., Study Chair — Hoosier Oncology Group, LLC; Nasser Hanna, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (7):
- United States (7):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - AP&S Clinic, Terre Haute, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Texas Oncology, PA, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Becerra CR, Hanna N, McCollum AD, Becharm N, Timmerman RD, DiMaio M, Kesler KA, Yu M, Yan T, Choy H. A phase II study with cetuximab and radiation therapy for patients with surgically resectable esophageal and GE junction carcinomas: Hoosier Oncology Group G05-92. J Thorac Oncol. 2013 Nov;8(11):1425-9. doi: 10.1097/JTO.0b013e3182a46c3b. PMID 24084441
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Assignment: Cetuximab 400 mg/m2 IV over 120 minutes Day -14 (Loading Dose) Cetuximab 250 mg/m2 IV over 60 minutes Day -7 Cetuximab 250 mg/m2 IV over 60 minutes Days 1, 8, 15, 22, 29 and 36
  Radiation Therapy: External beam radiation therapy, beginning on day 1, 4500 cGy to esophagus with boost of 540 cGy at 180 cGy per fraction for 6 weeks
  Surgery: Surgical resection of primary tumor and adjacent mediastinal and/or celiac lymph nodes by a transthoracic approach after satisfactory hematologic and functional recovery within 8 weeks of completion of radiation therapy
  Tissue Sample: For patients who give their consent, fresh frozen tissue will be obtained per EUS at baseline, per EUS 2 weeks after the initiation of chemotherapy, and at the time of surgery for pathology submission
Period: Overall Study
Arm/Group | Single Arm Assignment
Started | 41
Completed | 39
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 41
Age, Customized [Median (Full Range); unit: years]
  Median | 64 [50 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Tumor Site [Number; unit: participants]
  Esophagus | 26
  Gastroesophageal Junction | 15
Disease Stage [Number; unit: participants] — Stage I, Stage II, and Stage III Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV The cancer has spread to distant parts of the body.
  participants
    IIA | 10
    IIB | 7
    III | 22
    IVA | 2
Histology [Number; unit: participants]
  Squamous cell carcinoma | 9
  Adenocarcinoma | 32
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  participants
    0 | 26
    1 | 13
    2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathologic Response (pCR)
Description: To evaluate complete pathologic response rate in patients with esophageal and GE junction carcinomas.
  Complete pathologic response (pCR) is defined as the absence of tumor cells on the resected specimen in the esophagus and/or GE junction.
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Groups:
- Single Arm Assignment: Cetuximab 400 mg/m2 IV over 120 minutes Day -14 (Loading Dose) Cetuximab 250 mg/m2 IV over 60 minutes Day -7 Cetuximab 250 mg/m2 IV over 60 minutes Days 1, 8, 15, 22, 29 and 36 Combined with radiation therapy for six weeks. Surgical esophageal resection after 6 to 8 week rest period.
  Subjects who consent will provide tissue samples.
  Radiation Therapy: External beam radiation therapy, beginning on day 1, 4500 cGy to esophagus with boost of 540 cGy at 180 cGy per fraction for 6 weeks
  Surgery: Surgical resection of primary tumor and adjacent mediastinal and/or celiac lymph nodes by a transthoracic approach after satisfactory hematologic and functional recovery within 8 weeks of completion of radiation therapy
  Tissue Sample: For patients who give their consent, fresh frozen tissue will be obtained per EUS at baseline, per EUS 2 weeks after the initiation of chemotherapy, and at the time of surgery for pathology submission
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 39
percentage of participants | 36.6

2. Secondary Outcome: Complete Pathological Response Rate for Patients Who Underwent Esophagectomy.
Description: To evaluate complete pathologic response rate in patients with esophageal and GE junction carcinomas that underwent esophagectomy.
  Complete pathologic response (pCR) is defined as the absence of tumor cells on the resected specimen in the esophagus and/or GE junction.
Time Frame: Up to 36 months
Population: Participants who underwent esophagectomy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 31
percentage of participants
  Participants with a pCR | 48 [30 to 67]
  Participants with no pCR | 52 [33 to 70]

3. Secondary Outcome: Time to Relief of Dysphagia
Description: To evaluate time to relief of dysphagia in patients with esophageal and GE junction carcinomas receiving preoperative radiation and cetuximab
Time Frame: 36 months
Population: No data was collected or analyzed for this secondary objective.
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

4. Secondary Outcome: Evaluate Toxicity
Description: To evaluate the overall toxicities of preoperative radiation and cetuximab in patients with esophageal and GE junction carcinomas
Time Frame: 36 months
Population: Grade 3 toxicities occurring in >5% of participants are reported. Safety data is presented in totality in the adverse events section.
Measure: Number; unit: participants
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 41
participants
  Anorexia | 3
  Dehydration | 3
  Dyspagia | 7
  Dyspnea | 2
  Fatigue | 2
  Hypernatremia | 2

5. Secondary Outcome: Perform Exploratory Molecular Correlates.
Description: To perform exploratory molecular correlates to determine the mechanisms of response and resistance to cetuximab and radiation therapy.
Time Frame: 36 months
Population: No data was collected or analyzed for this secondary objective.
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

6. Secondary Outcome: Complete and Partial Response Rate for Patients by Disease Stage: IIA
Description: To evaluate complete and partial response rate of preoperative radiation and cetuximab in patients with esophageal and GE junction carcinomas
Time Frame: 36 months
Population: patients with IIA
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 10
percentage of participants | 70

7. Secondary Outcome: Complete and Partial Response Rate for Patients by Disease Stage: IIB
Description: as for outcome 6
Time Frame: 36 months
Population: patients with IIB
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 7
percentage of participants | 29

8. Secondary Outcome: Complete and Partial Response Rate for Patients by Disease Stage: III
Description: as for outcome 6
Time Frame: 36 months
Population: patients with Stage III disease
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 22
percentage of participants | 27

9. Secondary Outcome: Complete and Partial Response Rate for Patients by Histology: Adenocarcinoma
Description: as for outcome 6
Time Frame: 36 months
Population: patients with IIB
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 32
percentage of participants | 28

10. Secondary Outcome: Complete and Partial Response Rate for Patients by Histology: Squamous Cell
Description: as for outcome 6
Time Frame: 36 months
Population: patients with IIB
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 9
percentage of participants | 67

ADVERSE EVENTS:
Arm/Group | Single Arm Assignment
Serious Adverse Events (participants affected / at risk) | 16/41
Other Adverse Events (participants affected / at risk) | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Assignment (N=41)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (2)
BLOOD/BONE MARROW - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 1 (1)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 3 (4)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1)
FISTULA, GI / ESOPHAGUS (Gastrointestinal disorders) | 1 (1)
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 1 (1)
HEMORRHAGE, GI / ESOPHAGUS (Gastrointestinal disorders) | 1 (2)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / ABDOMEN NOS (Infections and infestations) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / CATHETER-RELATED (Infections and infestations) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1)
PAIN / BACK (General disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SODIUM, SERUM-HIGH (HYPERNATREMIA) (Investigations) | 2 (2)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 1 (1)
VASCULAR - OTHER (SPECIFY, __) (Vascular disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
WEIGHT LOSS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Assignment (N=41)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 2 (3)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 4 (4)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 2 (2)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 2 (2)
ANOREXIA (Gastrointestinal disorders) | 9 (15)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 2 (2)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 3 (4)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 5 (5)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (8)
DEHYDRATION (Gastrointestinal disorders) | 2 (2)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 5 (5)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 2 (2)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 35 (47)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ESOPHAGITIS (Gastrointestinal disorders) | 4 (6)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 15 (26)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 3 (3)
FLU-LIKE SYNDROME (General disorders) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 5 (6)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 2 (3)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 8 (9)
HEMOGLOBIN (Blood and lymphatic system disorders) | 3 (3)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (4)
HOT FLASHES/FLUSHES (Endocrine disorders) | 1 (1)
HYPERTENSION (Cardiac disorders) | 1 (1)
HYPOTENSION (Cardiac disorders) | 2 (2)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / CONJUNCTIVA (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / UPPER AIRWAY NOS (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 5 (5)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 1 (1)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 7 (11)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 4 (5)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 19 (24)
NEUROPATHY: SENSORY (Nervous system disorders) | 2 (2)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 3 (3)
PAIN / BACK (General disorders) | 2 (2)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PAIN / ESOPHAGUS (Gastrointestinal disorders) | 3 (3)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / FACE (General disorders) | 1 (1)
PAIN / HEAD/HEADACHE (General disorders) | 5 (6)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / PAIN NOS (General disorders) | 1 (1)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PAIN - OTHER (SPECIFY, __) (General disorders) | 5 (5)
PALPITATIONS (Cardiac disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 4 (5)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 14 (15)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 (1)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 31 (64)
RASH: DERMATITIS ASSOCIATED WITH RADIATION / CHEMORADIATION (Skin and subcutaneous tissue disorders) | 3 (3)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 3 (3)
RIGORS/CHILLS (General disorders) | 3 (3)
SEIZURE (Nervous system disorders) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (1)
STRICTURE/STENOSIS (INCLUDING ANASTOMOTIC), GI / ESOPHAGUS (Gastrointestinal disorders) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 6 (6)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
VOMITING (Gastrointestinal disorders) | 9 (16)
WEIGHT LOSS (General disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No